CLINICAL TRIAL: NCT07017010
Title: Optimizing Phonological Awareness Learning in Prekindergarten and Kindergarten to Improve Later Reading and Spelling
Acronym: Project OPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Florida State University (Other)
Responsible Party: Principal Investigator, Shayne B. Piasta, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OSUSTUDY20250377; R01HD112429 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-08

CONDITIONS: Reading Difficulties

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Dr. Schatschneider, who will have no role in recruitment/enrollment, no communication with participants/parents/teachers, and will be blind to children's pretest/screening assessment results, will randomly assign participating children within each center/school to study conditions. All child measures will be administered individually at the children's school by trained research assistants who are blind to the child's experimental condition to the extent possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- phonemic awareness intervention (PA) (Experimental): In the PA condition, children will receive 12 weeks of intervention, approximately 15 minutes per day, for 4 or 5 days per week, for a maximum of 48 lessons.
  Interventions: Behavioral: phonemic awareness intervention (PA)
- phonological sensitivity + phonemic awareness intervention (PSPA) (Experimental): In the PSPA condition, children will receive 12 weeks of intervention in 15- minute lessons, with a maximum of 48 lessons, 4 or 5 days per week.
  Interventions: Behavioral: phonological sensitivity + phonemic awareness intervention (PSPA)
- delayed onset phonemic awareness intervention (DPA) (Experimental): In the DPA condition, children will receive intervention that includes identical types of lessons to the PA condition but with a delayed onset to match the start of week 7 for other conditions. The difference will be that they receive instruction for only 6 weeks, or for a total of 24 maximum lessons. These also will be delivered for approximately 15 minutes each day, for 4 or 5 days per week.
  Interventions: Behavioral: delayed onset phonemic awareness intervention (DPA)
- Instruction-as-usual control (BAU) (No Intervention): In the BAU condition children will receive only their typical general education classroom instruction as provided by their classroom teacher. This will vary naturally from classroom to classroom.

INTERVENTIONS:
Behavioral: phonemic awareness intervention (PA) — All 12 weeks of lessons will exclusively focus on instruction at the phoneme level (i.e., the individual sounds in words), with activities addressing the blending of sounds to form short words. Other activities may include counting the number of sounds heard in a word, matching letter tiles to the sounds heard in the word, and separating short words into their component sounds.
  Arms: phonemic awareness intervention (PA)
Behavioral: phonological sensitivity + phonemic awareness intervention (PSPA) — The first six weeks of intervention will include a focus on being able to manipulate (separate and blend) parts of words larger than the individual sounds. This will include manipulating compound word components, syllables, and initial sounds and rhyming components of words. Activities may include matching pictures of words, assembling/disassembling puzzle pieces that represent words, and sorting pictures (words) by their first or ending sounds. The second six weeks of intervention will focus on phonemic awareness, as described for the PA intervention condition, and be the same as what the children in the DPA intervention condition experience.
  Arms: phonological sensitivity + phonemic awareness intervention (PSPA)
Behavioral: delayed onset phonemic awareness intervention (DPA) — The six weeks of intervention will focus on phonemic awareness, as described for the PA intervention condition, and be the same as the second six weeks of lessons that the children in the PSPA intervention condition experience.
  Arms: delayed onset phonemic awareness intervention (DPA)

SUMMARY:
The goal of the proposed study is to directly and rigorously address current scientific controversy about phonological awareness intervention content and timing for prekindergarten and kindergarten children. Using an experimental design, we will compare the relative impact of phonological sensitivity + phonemic awareness intervention versus phonemic awareness intervention on children's phonemic awareness and later reading and spelling abilities. We expect that both types of intervention will lead to impacts beyond business-as-usual instruction but do not have directional hypotheses as to which type of intervention will be most effective. Also, we will determine the relative efficacy of intervening in prekindergarten versus kindergarten, examine child characteristics that might moderate effects, and explore whether a transition point can be identified as to when phonemic awareness intervention may be most effective. Ultimately, our findings will help optimize early phonological awareness instruction.

ELIGIBILITY:
Inclusion Criteria:

* Parent consent
* Child assent
* Enrollment in prekindergarten or kindergarten
* At least 4 years old
* Score below the 50th percentile on the Phonological Awareness Component Score of the Comprehensive Test of Phonological Processing 2 (CTOPP 2).

Exclusion Criteria:

* Severe sensory impairment that interferes with the capacity to hear instructions or see visual stimuli as reported by parents on the initial Child/Family Survey.
* Inability to speak or understand English at a basic level, as indicated by a criterion score < 6 on the Clinical Evaluation of Language Fundamentals Preschool-3 Screening Test (CELF:PS).
* Severe behavior issues as indicated by (a) a score 3 on the aggressive behavior item of the externalizing subscale of the Student Risk Screening Scale-Early Childhood (SRSS-EC) or (b) a total score ≥ 16 on the externalizing subscale of the SRSS-EC.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Test of Preschool Early Literacy: PA subtest | screening/pretest (within first 3 months of school year prior to intervention), midtest (within 2 months following the first 6 weeks of intervention and before starting the second 6 weeks of intervention), posttest (within 3 months of intervention end)
  The TOPEL phonological awareness subtest includes 27 items with a focus on blending and deleting various sound components within words (e.g., compound word components, syllables, individual sounds). Some items do, and others do not include pictorial supports where children can respond by pointing to their answer.
Comprehensive Test of Phonological Processing 2: Elision, Blending Words, and Sound Matching subtests | screening/pretest (within first 3 mos, prior to intervention), midtest (within 2 mos after first 6 weeks of intervention, posttest (within 3 mos of intervention end), followup 1 (~15-18 mos after enrollment), followup 2 (PK only, ~27-30 mos after enroll)
  The CTOPP2 includes three core subtests that we will administer. Elision is a 34- item subtest to assess how participants can say a word then say what is left after leaving out designated sounds. Blending Words is a 33-item subtest to see how a participant would combine sounds by listening to a series of audio recorded separate sounds then putting together the sounds to make a full word. Sound matching is a 26-item subtest to see how a participant can match sounds. The examiner says a target word then says three other words while pointing to drawings showing the words. For the first 13 items, participants have to point to pictures that match the first sound in the target word and for the following 13 items they match the end sound.

SECONDARY OUTCOMES:
Woodcock-Johnson Tests of Achievement IV: Letter Word ID, Word Attack, and Spelling subtests | posttest (within 3 months of intervention end), followup 1 (~15-18 mos after enrollment), followup 2 (PK only, ~27-30 mos after enroll)
  We will administer three subtests of the widely used standardized measure the Woodcock-Johnson Tests of Achievement IV (WJ Letter Word ID, WJ Word Attack, and WJ Spelling). Letter Word ID requires children to correctly label individual letters and then individual words of increasing difficulty (maximum 75, with stopping rules after successive errors). Word Attack requires children to correctly pronounce nonwords of increasing length and difficulty (maximum 32, with stopping rules after successive errors). Spelling requires children to write the conventional spelling of words dictated to them by a recording (maximum 30, with stopping rules after successive errors).
Test of Word Reading Efficiency 2 | posttest (within 3 months of intervention end), followup 1 (~15-18 mos after enrollment), followup 2 (PK only, ~27-30 mos after enroll)
  The Test of Word Reading Efficiency 2 is a standardized and widely used measure of reading fluency. In both subtests children are given 45 seconds in which to read as many of a list of presented words as possible. In list one, the words are real words. In list two the words are pronounceable nonsense words. Both lists become increasingly difficult.
Word Spelling assessment | posttest (within 3 months of intervention end), followup 1 (~15-18 mos after enrollment), followup 2 (PK only, ~27-30 mos after enroll)
  The Word Spelling assessment includes two parts: asking children to spell 5 dictated real words and 5 dictated nonsense words, with each part scored separately.

CONTACTS AND LOCATIONS:
Overall Officials: Shayne B Piasta, PhD, Principal Investigator — Ohio State University; Beth M Phillips, PhD, Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The study will generate (a) longitudinal data concerning children's phonological awareness, reading and spelling, and other early literacy skills; (b) data concerning children's speech/language skills, working memory, and problem behavior at screening/pretest; and (c) descriptive data concerning child demographics, participating centers/schools, and intervention implementation/fidelity. We will share child behavioral data (raw scores plus normative scores when available), child demographic data (with age at first assessment rather than birthdate), center/school descriptive data, and summative scores for intervention implementation/fidelity data. We will make deidentified study data publicly available via LDbase. We will also use the Open Science Framework for sharing project protocols and analytic code, along with preregistrations for specific analyses related to main (or supplemental) aims.
Supporting Information: SAP, Analytic Code
Time Frame: Scientific data will be made available to other users no later than when we first publish findings addressing any of the specific aims or the end of the project period, whichever is sooner. Data will remain publicly available indefinitely via LDbase.
Access Criteria: Data will be publicly available and accessible via LDbase. Datasets posted in LDbase.com are reusable under a Creative Commons Attribution, Non-Commercial (CC-BY-NC) license. The data may be accessed by anyone for any types of analyses by downloading the datafiles from LDbase (i.e., there are no restrictions).
URL: https://doi.org/10.33009/ldbase.1744025400.0ceb

REFERENCES:
- See also: Project website — https://crane.osu.edu/our-work/project-optimizing-phonological-awareness-learning-opal/
- See also: Project Open Science Framework site — https://osf.io/9pynx/